CLINICAL TRIAL: NCT00498472
Title: NT-proBNP in the Optimization of Treatment After Recent Acute Heart Failure (BOT-AcuteHF) Trial
Brief Title: NT-proBNP in the Optimization of Treatment After Recent Acute Heart Failure Trial
Acronym: BOT_AcuteHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOT_1
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2007-07

CONDITIONS: Acute Heart Failure
Keywords: BNP; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Pre-discharge NT-ProBNP based
  Interventions: Procedure: Pre-discharge NT-ProBNP based treatment
- B (No Intervention): Discharge date and treatment not based on the knowledge of pre-discharge NT-proBNP levels

INTERVENTIONS:
Procedure: Pre-discharge NT-ProBNP based treatment — Discharge date, treatment and follow-up based also on the knowledge of NT-ProBNP levels measured at 2-3 days before discharge.
  Discharge may be postponed and medical treatment may be changed when NT-ProBNP is >3000 pg/ml. Changes in medical treatment will include the following: increase in the diuretic dose, association of a different diuretic; combination of digoxin therapy; increase in the dose of the renin-angiotensin inhibitor; association of an ARB; association of a nitrate; short course of i.v. diuretic, vasodilator and/or inotropic therapy.
  Arms: A

SUMMARY:
Hospitalizations for acute heart failure syndromes (AHFS) are associated with a high rehospitalisation and mortality rate. The aim of this study is to assess if the measurement of NT-proBNP levels before discharge may improve the prognosis of the patients recently admitted to hospital for AHFS

DETAILED DESCRIPTION:
Study population. We will include into the study patients admitted to our institute for AHFS with New York Heart Association (NYHA) class III or IV symptoms. All patients should have evidence of symptomatic heart failure with symptoms at rest or during minimal exercise requiring intravenous therapy.

All patients should give their written informed consent before entry into the study. Patients with clinical or laboratory evidence of an acute coronary syndrome as well as patients with major arrhythmias will be excluded if these conditions are likely to be the main cause of the symptoms. In contrast, patients with aspecific electrocardiographic ST segment changes and/or with a slight elevation of plasma troponin levels may be included as these conditions are known to be frequently associated with AHFS and it is generally not possible to establish to which extent they are the cause rather than the consequence of the hemodynamic decompensation. The patients in whom a coronary revascularization procedure (either PTCA or CABG) is planned in the next 3 months and the patients with non cardiac concomitant diseases that may influence outcome as primary factor will be excluded from the study.

Study design. Blood samples for the assessment of NT-proBNP plasma levels will be obtained in all the patients at at least two time intervals: pre-discharge (e.g. 24 to 72 hours before the planned date of discharge) and at discharge (e.g. at the day of discharge). Pre-discharge samples will be taken when the patient is clinically stable, on the same oral drugs and at the same doses which are planned to be administered after discharge.

All patients will be randomised according to a previous randomization scheme to two groups: control group, in which the results of NT-proBNP levels will be known only retrospectively, at the end of the trial; intervention group, in which the values of pre-discharge NT-proBNP plasma levels will be known by the investigator on the day after that of the blood sample.

In the intervention group, it will be possible to change medical treatment and, if needed, prolong the hospitalization, in the case that the pre-discharge NT-proBNP levels are >3000 pg/mL. This value has been associated with a 13-fold increase in mortality and heart failure rehospitalisation rates in patients recently admitted for AHFS. (Eur J Heart Fail. 2007 Jun 15; [Epub ahead of print] PMID: 17573240) The following changes of treatment will be possible: increase in the dose of the diuretic, association of a different diuretic (e.g. an aldosterone antagonist); combination of digoxin therapy; increase in the dose of the rennin-angiotensin inhibitor; association of an angiotensin receptor blocker; association of a nitrate; short course of i.v. diuretic, vasodilator and/or inotropic therapy.

Plasma levels of NT-proBNP will then be measured at discharge. It is our aim to use in the intervention group a treatment modality similar to that which may be expected if NT-proBNP levels are used to guide therapy. Therefore, the clinical investigator assessing these patients may require to the laboratory knowledge of the discharge NT-proBNP levels and delay patient's discharge and further adjust treatment, in case that the response to treatment (e.g. the decrease in NT-proBNP levels) be found as insufficient.

In the intervention group, a further assessment of plasma NT-proBNP levels will be repeated 7 to 21 days after discharge. If the NT-propBNP levels will still be elevated at that time, the investigator may further change medical treatment.

A satisfactory change in NT-ProBNP plasma levels is defined a priori as either one of the following: a) a decrease in plasma NT-proBNP below 3000 pg/mL (a value which has been associated with a favourable prognosis in our previous study group); b) a decrease > 30% from the first values detected (i.e. those measured 24 to 72 hours before discharge). This percentage is based on previous studies regarding both the prognostic value of serial changes in NT-proBNP levels and their spontaneous week to week variability in clinically stable heart failure patients.

Additional exams. During the hospitalization, all patients will have at least daily assessments of their clinical conditions with medical treatment titrated to obtain clinical stability and symptoms relief, if possible. The investigator will be unaware of the randomization code until the day of the pre-discharge sample. No differences in baseline clinical characteristics, hospitalization duration before the planned discharge and in-hospital treatment are expected between the two study groups.

All the patients will undergo a standard Doppler-echocardiography and chest-X ray at least once during the hospitalization. The 6 minutes walk distance will be measured when the patient will be clinically stable, before discharge.

Follow-up. Each patient will undergo a clinical visit or a telephone assessment of his/her clinical conditions at 1 and 3 months after discharge and every 6 months thereafter until the end of the study. Unplanned ambulatory visits will be allowed based on the clinical conditions and needs of the patient. An echocardiographic exam and the assessment of the 6 minutes walk distance will be repeated 6 months after the initial hospitalization. Standard laboratory exams will be repeated at 1, 3 and 6 months after discharge

Outcome measures Main outcome: Incidence of unplanned cardiovascular hospitalization and cardiac deaths at 6 months in the control and the intervention groups.

Secondary outcomes: Incidence of cardiac mortality alone; combined incidence of cardiac deaths, cardiovascular hospitalizations and unplanned ambulatory visits; number of days spent in hospital during the first hospitalization; number of days spent in the hospital during follow-up; changes in the left ventricular ejection fraction, volumes and filling patterns from the first hospitalization to after 6 months; changes in NYHA class and in 6 minutes walk distance; changes in renal function from baseline to discharge and from discharge to the reassessment at 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for acute HF with New York Heart Association class III or IV symptoms.
* Requirement of intravenous therapy
* All patients should give their written informed consent

Exclusion Criteria:

* Clinical or laboratory evidence of an acute coronary syndrome
* Major arrhythmias as main cause of symptoms
* Patients in whom a coronary revascularization procedure (either PTCA or CABG) is planned in the next 3 months
* Non cardiac concomitant diseases which may have an important influence on outcome as primary factor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2006-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Incidence of unplanned cardiovascular hospitalization and cardiac deaths at 6 months in the control and the intervention groups. | 30 months

SECONDARY OUTCOMES:
Cardiac mortality alone | 30 months
Combined end-point of cardiac deaths, cardiovascular hospitalizations; no. of days in hospital during follow-up | 30 months
Changes in LVEF, LV volumes, 6MWTD, NYHA class from discharge to 6 mts. f-up | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Metra, MD, Principal Investigator — Section of Cardiovascular Disease, University of Brescia
Locations (1):
- Cardiologia, University of Brescia c/o Spedali Civili P.zza Spedali Civili 1, Brescia, BS, Italy

REFERENCES:
- [Background] Metra M, Nodari S, Parrinello G, Specchia C, Brentana L, Rocca P, Fracassi F, Bordonali T, Milani P, Danesi R, Verzura G, Chiari E, Dei Cas L. The role of plasma biomarkers in acute heart failure. Serial changes and independent prognostic value of NT-proBNP and cardiac troponin-T. Eur J Heart Fail. 2007 Aug;9(8):776-86. doi: 10.1016/j.ejheart.2007.05.007. Epub 2007 Jun 18. PMID 17573240
- [Background] Bettencourt P, Azevedo A, Pimenta J, Frioes F, Ferreira S, Ferreira A. N-terminal-pro-brain natriuretic peptide predicts outcome after hospital discharge in heart failure patients. Circulation. 2004 Oct 12;110(15):2168-74. doi: 10.1161/01.CIR.0000144310.04433.BE. Epub 2004 Sep 27. PMID 15451800